CLINICAL TRIAL: NCT01161251
Title: Atrial Fibrillation Registry for Ankle-brachial Index Prevalence Assessment: Collaborative Italian Study.
Acronym: ARAPACIS
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Prof., University of Roma La Sapienza
Other Study IDs: SIMI-ARA PACIS
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Atrial Fibrillation; Peripheral Vascular Disease
Keywords: Atrial Fibrillation; ABI; PAD; Registry; Italian
MeSH Terms: conditions — Atrial Fibrillation; Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Atrial fibrillation patients: Non-valvular atrial fibrillation (paroxysmal, persistent or permanent)

SUMMARY:
Atrial fibrillation (AF) is the most common sustained dysrhythmia encountered in clinical practice in North America and Europe, accounting for approximately one-third of all hospitalizations for a cardiac rhythm abnormality. The presence of AF markedly increases the patient's risk for developing arterial embolism and stroke, depending on the presence of other clinical conditions, such as hypertension and diabetes. AF is associated with a fivefold increased risk for stroke, and is estimated to cause 15% of all strokes.

Patients with AF frequently have several risk factors for atherosclerosis, including hypertension, diabetes, and dyslipidemia. Accordingly, systemic signs of atherosclerosis can be detected in AF patients, and these likely accounts for an enhanced risk of coronary heart disease. In addition to cerebrovascular disease, patients with AF may suffer from coronary events including myocardial infarction (MI), but the rate of MI in AF patients seems to be variable, but often underestimated.

Moreover, coexistence of peripheral arterial disease (PAD) is a relevant clinical sign of systemic atherosclerosis.

Ankle-brachial index (ABI) is a simple, inexpensive, and non-invasive PAD measurement, even at the pre-symptomatic phase when intervention can improve prognosis and prevent or delay severe complications ABI is calculated by measuring the systolic blood pressure in the posterior tibial and/or the dorsalis pedis arteries either in both legs or 1 leg chosen at random (using a Doppler probe or alternative pulse sensor), with the lowest ankle pressure then divided by the brachial systolic blood pressure. In addition to peripheral artery disease, the ABI also is an indicator of generalized atherosclerosis because lower levels have been associated with higher rates of concomitant coronary and cerebrovascular disease, and with the presence of cardiovascular risk factors.

Two large studies in patients with AF document the existence of PAD in about 3-5% of patients. It is possible, however, that such an incidence has been underestimated as only symptomatic patients were considered as affected by PAD. As PAD is an important marker of systemic atherosclerosis, its association with AF reinforces the concept that patients with AF have systemic atherosclerosis that potentially account for coronary complications.

To date, a national registry of AF patients is not available to verify the real impact of cardiovascular events in this clinical setting.

DETAILED DESCRIPTION:
Study design: Prospective longitudinal study

Methods and Materials: The investigators planned to assess at baseline and at scheduled follow up visits :

1. Ankle-Brachial Index measurement
2. Anamnestic clinical information and Anthropometric measurements
3. Echocardiogram (volume size), electrocardiogram (AF type)
4. Outcome events such as nonfatal or fatal acute myocardial infarction, target lesion or vessel revascularization nonfatal or fatal ischemic stroke, transient ischemic attack, death from any cardiac or vascular cause, death from any cause Study duration: 3 years follow-up Statistical methods: The prevalence will be calculated by exact confidence intervals (Wilson method). The cumulative incidence will be calculated by the product-limit estimator of Kaplan-Meyer and presented with confidence intervals at 95%. The incidences and prevalences will be then adjusted through appropriate multivariate analysis (using the Cox proportional hazards model and logistic model) that will take into account the effect of potential confounders. Similarly, the effect-center presence will be checked and possibly removed. Secondary endpoints will be assessed by using Log-rank test method, and by the Cox model (with time-dependent effects) multivariate analysis.

Subgroups analysis will be also conducted for patients with first onset of AF or recurrent AF Sample size: The investigators plan to include in the study n = 3,000 AF patients, with competitive recruitment between centers involved in the study. The sample size was calculated assuming an expected prevalence of 19% at time zero, and in order to obtain a confidence interval 95% to prevail at time zero whose distance from the edge is less than or equal to 1.4%. This sample size yields a power greater than 99.9% for the secondary endpoint, assuming an event rate of 19% for patients with ABI <=0.9, and 10% for patients with ABI >0.9.An interim analysis showed an ABI prevalence, calculated by exact confidence intervals, of 21% in patients with AF, it is considered to interrupt the enrollment, as the observed prevalence is greater than two percentage points higher than that assumed. The sample size is amended as follows: a sample of 2027 patients leads to the expected prevalence of 21% with a confidence interval width of 3.5. This sample size has no impact on the power of the secondary objective.

ELIGIBILITY:
Inclusion Criteria:

* Non-valvular atrial fibrillation (paroxysmal, persistent or permanent)
* Genders Eligible for Study: Both
* Ages Eligible for Study 18 years and older
* Signed written informed consent

Exclusion Criteria:

* Valvular AF
* Cancer
* Disease with life expectancy less than 3 years
* Pregnancy
* Hyperthyroidism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to include in the study n = 3,000 AF patients, with competitive recruitment between centers involved in the study. The sample size was calculated assuming an expected prevalence of 19% at time zero, and in order to obtain a confidence interval 95% to prevail at time zero whose distance from the edge is less than or equal to 1.4%. This sample size yields a power greater than 99.9% for the secondary endpoint, assuming an event rate of 19% for patients with ABI <=0.9, and 10% for patients with ABI >0.9.An interim analysis showed an ABI prevalence, calculated by exact confidence intervals, of 21% in patients with AF, it is considered to interrupt the enrollment, as the observed prevalence is greater than two percentage points higher than that assumed. The sample size is amended as follows: a sample of 2,027 patients leads to the expected prevalence of 21% with a confidence interval width of 3.5. This sample size has no impact on the power of the secondary objective.
Sampling Method: Probability Sample
Enrollment: 2027 (Actual)
Dates: Start 2010-07; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
ABI PREVALENCE | 1 year
  To estimate peripheral artery disease prevalence (defined by an Ankle-brachial index <=0.9) in AF patients.

SECONDARY OUTCOMES:
Vascular Events | 3 years
  To Estimate ischemic cardiovascular and cerebro-vascular events (fatal or non-fatal ) incidence in AF patients with or without peripheral artery disease

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, Full Prof, Study Chair — Prima Clinica Medica - Sapienza University of Rome
Locations (2):
- Italy (2):
  - Sapienza - University of Rome and SIMI, Rome, Italy
  - Società Italiana di Medicina Interna, Rome, Rome

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Mannucci PM, Nobili A. Appropriateness of antithrombotic prophylaxis in the oldest old with non-valvular atrial fibrillation: ARAPACIS and REPOSI. Eur J Intern Med. 2015 Nov;26(9):e47-8. doi: 10.1016/j.ejim.2015.08.013. Epub 2015 Sep 5. No abstract available. PMID 26350113
- [Background] Pignatelli P, Pastori D, Perticone F, Corazza GR, Violi F; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) Study group. Lights and shadows in the management of old and new oral anticoagulants in the real world of atrial fibrillation by Italian internists. A survey from the Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study. Eur J Intern Med. 2015 Oct;26(8):e31-3. doi: 10.1016/j.ejim.2015.06.007. Epub 2015 Jun 27. No abstract available. PMID 26123820
- [Background] Violi F, Pastori D, Perticone F, Hiatt WR, Sciacqua A, Basili S, Proietti M, Corazza GR, Lip GY, Pignatelli P; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) STUDY group. Relationship between low Ankle-Brachial Index and rapid renal function decline in patients with atrial fibrillation: a prospective multicentre cohort study. BMJ Open. 2015 May 21;5(5):e008026. doi: 10.1136/bmjopen-2015-008026. PMID 25998039
- [Result] Violi F, Davi G, Proietti M, Pastori D, Hiatt WR, Corazza GR, Perticone F, Pignatelli P, Farcomeni A, Vestri AR, Lip GY, Basili S; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) STUDY Investigators. Ankle-Brachial Index and cardiovascular events in atrial fibrillation. The ARAPACIS Study. Thromb Haemost. 2016 Apr;115(4):856-63. doi: 10.1160/TH15-07-0612. Epub 2016 Jan 7. PMID 26740316
- [Result] Proietti M, Marra AM, Tassone EJ, De Vuono S, Corrao S, Gobbi P, Perticone F, Corazza GR, Basili S, Lip GY, Violi F, Raparelli V; ARAPACIS Study Investigators; GIS Group. Frequency of Left Ventricular Hypertrophy in Non-Valvular Atrial Fibrillation. Am J Cardiol. 2015 Sep 15;116(6):877-82. doi: 10.1016/j.amjcard.2015.05.060. Epub 2015 Jun 25. PMID 26183791
- [Result] Proietti M, Calvieri C, Malatino L, Signorelli S, Corazza GR, Perticone F, Vestri AR, Loffredo L, Davi G, Violi F, Basili S; ARAPACIS (Atrial Fibrillation Registry for Ankle-Brachial Index Prevalence Assessment-Collaborative Italian Study) STUDY Investigators. Relationship between carotid intima-media thickness and non valvular atrial fibrillation type. Atherosclerosis. 2015 Feb;238(2):350-5. doi: 10.1016/j.atherosclerosis.2014.12.022. Epub 2014 Dec 20. PMID 25555267
- [Result] Raparelli V, Proietti M, Butta C, Di Giosia P, Sirico D, Gobbi P, Corrao S, Davi G, Vestri AR, Perticone F, Corazza GR, Violi F, Basili S; ARAPACIS Study Investigators; GIS Group. Erratum to: medication prescription and adherence disparities in non valvular atrial fibrillation patients: an Italian portrait from the ARAPACIS study. Intern Emerg Med. 2015 Mar;10(2):261-5. doi: 10.1007/s11739-014-1166-4. No abstract available. PMID 25519853
- [Result] Raparelli V, Proietti M, Butta C, Di Giosia P, Sirico D, Gobbi P, Corrao S, Davi G, Vestri AR, Perticone F, Corazza GR, Violi F, Basili S. Medication prescription and adherence disparities in non valvular atrial fibrillation patients: an Italian portrait from the ARAPACIS study. Intern Emerg Med. 2014 Dec;9(8):861-70. doi: 10.1007/s11739-014-1096-1. Epub 2014 Jul 3. PMID 24990547
- [Result] Violi F, Davi G, Hiatt W, Lip GY, Corazza GR, Perticone F, Proietti M, Pignatelli P, Vestri AR, Basili S; ARAPACIS Study Investigators. Reply: ankle-brachial index in patients with nonvalvular atrial fibrillation. J Am Coll Cardiol. 2014 Apr 15;63(14):1457-8. doi: 10.1016/j.jacc.2013.11.011. Epub 2013 Dec 4. No abstract available. PMID 24315905
- [Result] Violi F, Davi G, Hiatt W, Lip GY, Corazza GR, Perticone F, Proietti M, Pignatelli P, Vestri AR, Basili S; ARAPACIS Study Investigators. Prevalence of peripheral artery disease by abnormal ankle-brachial index in atrial fibrillation: implications for risk and therapy. J Am Coll Cardiol. 2013 Dec 10;62(23):2255-6. doi: 10.1016/j.jacc.2013.07.035. Epub 2013 Aug 14. No abstract available. PMID 23954332
- See also: Società Italiana di Medicina Interna — http://www.simi.it/